CLINICAL TRIAL: NCT01594021
Title: Efficacy of Preemptive Volume Loading to Prevent Arterial Hypotension During Induction of General Anesthesia
Acronym: NICOM-MAP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty of realization of the study
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/13; 2012-A00368-35 (Other: ANSM)
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia
Keywords: propofol; anesthesia, induction; hypotension; cardiac output
MeSH Terms: conditions — Hypotension | interventions — Gelatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High pre-emptive volume loading (Experimental)
  Interventions: Drug: Gelatin 500 mL
- Low pre-emptive volume loading (Active Comparator)
  Interventions: Drug: Gelatin 50 mL

INTERVENTIONS:
Drug: Gelatin 500 mL — intravenous administration
  Arms: High pre-emptive volume loading
Drug: Gelatin 50 mL — intravenous administration
  Arms: Low pre-emptive volume loading

SUMMARY:
Induction of general anesthesia induces frequently arterial hypotension. The short term goal of this study is to evaluate if preemptive volume loading prevents such complication.

DETAILED DESCRIPTION:
This is a randomized, prospective study which will include a total of 200 patients who are scheduled to undergo elective surgery. The research participants will be randomly assigned to

* a control group that will receive a low preemptive volume loading (50 mL of gelatin),
* a protocol group that will receive a high preemptive volume loading (500 mL of gelatin).

Volume loading is preceded by the measurement of stroke volume and cardiac output before and after a passive leg elevation test and followed by a standardized anesthetic protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective surgery.

Exclusion Criteria:

* Difficult peripheral venous access
* Allergy to gelatin
* Symptomatic cardiac disease, rhythm trouble, pace-maker, aortic valvular disease, aortic disease
* Morbid obesity, low BMI,
* hypovolemia,
* Raynaud syndrome or scleroderma,
* Contra-indication to propofol, remifentanil or to the use of Bispectral Index,
* Hematocrit < 20%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hypotension | 30 minutes
  mean arterial pressure less than 70% of the baseline measurement

SECONDARY OUTCOMES:
hemodynamic effect of leg passive elevation test | 30 minutes
hemodynamic effect of volume loading | 30 minutes
heart rate monitoring | 30 minutes
propofol dose when bispectral index is 50 | 30 minutes
propofol site effect concentration when bispectral index is 50 | 30 minutes
arterial pressure monitoring | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, Principal Investigator — Hopital Foch; Marc Fischler, Study Director — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France